CLINICAL TRIAL: NCT01984047
Title: A Phase 1, Randomized, Double-Blind (Sponsor Open), Placebo-Controlled, Single Dose Escalation Trial to Evaluate the Safety, Tolerability Pharmacokinetics and Pharmacodynamics of GSK3050002 (Anti-CCL20 Monoclonal Antibody) in Healthy Male Volunteers
Brief Title: Single Dose Escalation Trial to Evaluate the Safety, Tolerability Pharmacokinetics and Pharmacodynamics of GSK3050002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 200784
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Colitis, Ulcerative
Keywords: safety; GSK3050002; CCR6 receptor; single dose escalation; Phase 1; CCL20
MeSH Terms: conditions — Colitis, Ulcerative | interventions — GSK3050002

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- GSK3050002 0.1 mg (Experimental): Six subjects in this cohort will receive a single dose of GSK3050002 0.1 mg and two subjects will receive a single dose of placebo intravenously. Sentinel subjects (i.e. 1 subject will be dosed with GSK3050002 and 1 with placebo before the remainder of the cohort is dosed) will be used in the cohort.
  Interventions: Drug: GSK3050002; Drug: Placebo
- GSK3050002 0.5 mg (Experimental): Six subjects in this cohort will receive a single dose of GSK3050002 0.5 mg and two subjects will receive a single dose of placebo intravenously. Sentinel subjects will be used in the cohort.
  Interventions: Drug: GSK3050002; Drug: Placebo
- GSK3050002 1 mg (Experimental): Six subjects in this cohort will receive a single dose of GSK3050002 1 mg and two subjects will receive a single dose of placebo intravenously. Sentinel subjects will be used in the cohort
  Interventions: Drug: GSK3050002; Drug: Placebo
- GSK3050002 5 mg (Experimental): Six subjects in this cohort will receive a single dose of GSK3050002 5 mg and two subjects will receive a single dose of placebo intravenously. Sentinel subjects will be used in the cohort.
  Interventions: Drug: GSK3050002; Drug: Placebo
- GSK3050002 10 mg (Experimental): Six subjects in this cohort will receive a single dose of GSK3050002 10 mg and two subjects will receive a single dose of placebo intravenously. Sentinel subjects will be used in the cohort.
  Interventions: Drug: GSK3050002; Drug: Placebo
- GSK3050002 20 mg (Experimental): Six subjects in this cohort will receive a single dose of GSK3050002 20 mg and two subjects will receive a single dose of placebo intravenously. Sentinel subjects will be used in the cohort.
  Interventions: Drug: GSK3050002; Drug: Placebo

INTERVENTIONS:
Drug: GSK3050002 — GSK3050002 is a white to off-white lyophilized powder that will be reconstituted with sterile water for intravenous infusion. It is available in the concentrations of 0.1 milligram (mg)/kg, 0.5 mg/kg, 1 mg/kg, 5 mg/kg, 10 mg/kg and 20 mg/kg.
Drug: Placebo — Placebo contains normal saline (0.9% sodium chloride) for intravenous infusion

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of GSK3050002 in humans. Subjects will attend the clinical unit for a screening visit and if eligible and consenting, will attend to participate in the study within 30 days. Subjects will be admitted to the clinical unit the evening prior to dosing when each subject will receive a single intravenous dose of GSK3050002 or placebo, then remain in house under supervision until discharged on Day 3. Subjects will then return for 7 outpatient visits scheduled over the following 81 days. Finally, the follow-up visit will be 7-14 days following the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Male aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and 12- lead ECG. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria may be included only if the Investigator in consultation with the GSK Medical Monitor [if required] agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body mass index (BMI) within the range 18 - 29 kilogram per meter square [kg/m^2] (inclusive).
* Male subjects with female partners of child-bearing potential must agree to use one of the listed contraception methods. This criterion must be followed for 1 month prior to the first dose of study medication for 15 weeks post dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Suitable for cannulation and with adequate venous access.
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <= 1.5xUpper limit of Normal [ULN] (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on a single ECG QTcF < 450 milliseconds (msec).

Exclusion Criteria:

* Criteria Based Upon Medical Histories
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of severe drug allergies including type 1 hypersensitivity reaction to parental administration of contrast agents, human or murine proteins or monoclonal antibodies.
* Subject has acne which requires prescription treatment
* Criteria Based Upon Diagnostic Assessments
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for Human immunodeficiency virus (HIV) antibody.
* Subject is a heavy smoker as defined by a positive smoking breath test of >10 parts per million (ppm) carbon monoxide (CO).
* Other Criteria
* Evidence of current or at risk of developing bacterial, fungal, or viral infection at screening or within 7 days before dosing.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Subject is unable to refrain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements), within 7 days prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study.
* Subject is unable to abstain from travelling to area which carry a high risk of infection for the duration of the study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Subject is unable to abstain from being vaccinated or immunized for 4 weeks prior to dosing and for 19 weeks after the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2015-02-23 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Up to Day 98
  Adverse events will be collected from the start of study treatment until the follow-up contact
Laboratory measurements | Up to Day 98
  Clinical laboratory assessments will include haematology, clinical chemistry, urinalysis and other screening tests
Electrocardiogram (ECG) assessment as a measure of safety | Up to Day 98
  Triplicate 12-lead ECG will be recorded before dosing on Day 1 (Pre-dose) and a single 12-lead ECG will be obtained at all other timepoints
Vital signs as a measure of safety | Up to Day 98
  Vital sign measurements will include systolic and diastolic blood pressure, temperature, and pulse rate
Pharmacokinetic (PK) parameters after a single intravenous dose of GSK3050002 | Day 1, Day 2, Day 3, Day 7, Day 14, Day 21, Day 28, Day 42, Day 56 and Day 84
  The following PK parameters will be determined: maximum observed serum concentration (Cmax), time to Cmax (tmax), area under the serum concentration-time curve (AUC[0-t] and AUC[0-infinity]), and apparent terminal phase half-life (t1/2)

SECONDARY OUTCOMES:
Chemokine (C-C motif) ligand 20 (CCL20) levels in blood | Up to Day 87
  Whole blood may be collected for in vitro stimulation and measurement of CCL20 activity in a biological assay. Analysis of serum levels of total (free and drug bound) CCL20 may be performed
Immunogenicity development as assessed from anti-drug antibody | Up to Day 87
  An assay for detecting anti-drug antibodies (ADA) against GSK305002 will be developed and validated using an electrochemiluminescent (ECL) bridging assay. Testing will be performed using the typical tiered approach involving screening, confirmation, and titration assays. If sera contain potential anti- GSK3050002 antibodies, they will be confirmed by immunocompetition using excess drug. Confirmed samples with such antibodies will be further analyzed for titers and may be characterized for neutralizing activity by a neutralization assay

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Laffan SB, Thomson AS, Mai S, Fishman C, Kambara T, Nistala K, Raymond JT, Chen S, Ramani T, Pageon L, Polsky R, Watkins M, Ottolangui G, White JR, Maier C, Herdman M, Bouma G. Immune complex disease in a chronic monkey study with a humanised, therapeutic antibody against CCL20 is associated with complement-containing drug aggregates. PLoS One. 2020 Apr 23;15(4):e0231655. doi: 10.1371/journal.pone.0231655. eCollection 2020. PMID 32325480
- See also: Results for study 200784 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200784?search=study&study_ids=200784#rs